CLINICAL TRIAL: NCT07074106
Title: DespaTIL Study: A Phase II Trial of De-escalated Neoadjuvant Chemotherapy for Early-Stage Triple-Negative Breast Cancer Guided by Tumor-Infiltrating Lymphocytes (TILs) and Radiologic Response
Brief Title: TIL-Driven De-escalated Chemotherapy in Stage I-II TNBC
Acronym: DespaTIL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Grupo Brasileiro de Estudos do Câncer de Mama (GBECAM) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 831-25-ONCOLOGIA-IDOR-SP-M-I
Record Dates: First submitted 2025-07-09; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: TILs; Breast cancer; radiological response; Descalonation of neoadjuvant treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carboplatin and Taxane - 4 Cycles (Experimental): All patients will receive Carboplatin and a Taxane for 4 cycles. Patients who achieve a complete radiological response will proceed directly to surgery. Those without a complete radiological response will receive Doxorubicin and Cyclophosphamide, with or without Pembrolizumab, for an additional 4 cycles before surgery.
  Interventions: Drug: Carboplatin and a Taxane

INTERVENTIONS:
Drug: Carboplatin and a Taxane — All patients will receive Carboplatin and a Taxane for 4 cycles.
  * Patients who achieve a complete radiological response will proceed directly to surgery.
  * Patients without a complete radiological response will receive Doxorubicin and Cyclophosphamide, with or without Pembrolizumab, for an additional 4 cycles before surgery.

SUMMARY:
This is a phase II clinical study testing a more personalized and lighter chemotherapy approach for women with stage I or II triple-negative breast cancer. The treatment is adjusted based on signs from the immune system (called tumor-infiltrating lymphocytes, or TILs) and imaging results during treatment.

Patients with stage I triple-negative breast cancer (regardless of TIL levels) and those with stage II disease and high TILs (50% or more) will receive a combination of two chemotherapy drugs (carboplatin and a taxane) for four cycles.

If imaging shows the tumor has completely disappeared after this treatment, the patient will go straight to surgery. If the tumor is still visible, the treatment will be strengthened with additional chemotherapy drugs (anthracycline and cyclophosphamide), with or without a medicine called pembrolizumab, which helps the immune system fight cancer.

The main goal of the study is to see how many patients have a complete disappearance of the cancer after treatment. Other goals include understanding how imaging results relate to what is found during surgery and tracking how long patients live without the cancer coming back.

DETAILED DESCRIPTION:
This is a phase II, single-arm clinical trial investigating a de-escalated neoadjuvant chemotherapy regimen for stage I and II triple-negative breast cancer (TNBC), guided by tumor-infiltrating lymphocytes (TILs) and radiologic response.

Patients with stage I TNBC (regardless of TIL levels) and stage II TNBC with TILs ≥ 50% will receive four cycles of carboplatin and a taxane. Those who achieve a complete radiologic response will proceed to surgery, while patients without a complete radiologic response will be escalated to a regimen including anthracycline and cyclophosphamide, with or without pembrolizumab.

The primary objective is to evaluate the pathological complete response rate. Secondary outcomes include the correlation between radiologic and pathologic response, event-free survival, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary invasive breast carcinoma.
* One of the following conditions:
* Clinical stage T1c N0 M0 with any level of TILs; or
* Clinical stage T2 N0 M0 with TILs ≥ 50%.
* Estrogen receptor (ER) and progesterone receptor (PR) expression < 10%.
* HER2-negative or non-amplified, according to current ASCO-CAP criteria.
* No evidence of distant metastasis based on imaging performed prior to study entry (chest/abdomen/pelvis CT scan or FDG PET-CT).
* Age ≥ 18 years.
* ECOG performance status of 0 to 2.
* Adequate organ function

Exclusion Criteria:

* The subject has an uncontrolled severe concomitant condition, including but not limited to: active or ongoing infection, unstable angina, uncontrolled cardiac arrhythmia, congestive heart failure (NYHA Class III or IV), active ischemic heart disease, or chronic liver or kidney disease.
* Pregnant or breastfeeding participants.
* History of severe allergic reactions, including anaphylaxis or other hypersensitivity reactions to platinum-based agents or taxanes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate after 4 cycles of Carboplatin plus Paclitaxel. | 3 mo

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Instituto D'Or de Pesquisa e Ensino de Brasília, Brasília
  - Instituto D'Or de Pesquisa e Ensino de Curitiba, Curitiba
  - Instituto D'Or de Pesquisa e Ensino do Rio de Janeiro, Rio de Janeiro
  - Instituto D'Or de Pesquisa e Ensino de Salvador, Salvador
  - Instituto D'Or de Pesquisa e Ensino de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No